CLINICAL TRIAL: NCT03550300
Title: Muscle MRI in Charcot Mary Tooth Disease: a Prospective Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: University of Iowa (Other)
Responsible Party: Sponsor
Other Study IDs: 18/0244
Record Dates: First submitted 2018-05-14; First posted 2018-06-08 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-05

CONDITIONS: Charcot-Marie-Tooth Disease, Type IA; Charcot-Marie-Tooth Disease Type 2A; Charcot-Marie-Tooth Disease, Type IB; Charcot-Marie-Tooth Disease, Type X
MeSH Terms: conditions — Charcot-Marie-Tooth Disease; Charcot-Marie-Tooth disease, Type 2A; Charcot-Marie-Tooth disease, X-linked, 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for plasma NEFL levels will be optional at both research visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with CMT: Participants with CMT1A, CMT1B, CMT2A or CMTX1
- Control participants: Control participants

SUMMARY:
This cohort study (participants with CMT and control participants) has two parts (Part 1: CMT1A cohort; Part2: CMT1B, CMT2A and CMTX1 cohort) and is proposed to take place over 3 years across three sites. Participants with CMT aged 5-60 for potential enrolment in the trial will be identified through the existing inherited neuropathy clinics at each site and control participants will be identified among the unaffected relatives and carers of the participants with CMT. If they show interest in participating, they will be given the relevant Patient Information Sheets, Written Consent forms and/or Assent forms. Half of the participants will be recruited at the UK sites (NHNN and GOSH) and the other half at the US collaborating site. Each participant will be invited to two separate research visits (12 months apart) for which travel expenses (return journey) will be reimbursed. Each research visit is expected to last approximately 3 hours and during it, relevant detailed clinical data will be collected (CMTPedS for participants with CMT aged 5-20, CMTESv2-R for participants with CMT over the age of 10, CMT-HI for participants with CMT over the age of 16) and the participant will also undergo an MRI scan (up to 45 minutes) of the lower limbs (feet and calves or calves and thighs). Two separate neuromuscular MRI protocols with specific sequences will be used for the scans of foot and calf muscles and scans of calf and thigh muscles. Blood samples for plasma NEFL levels will be optional at both research visits for the participants at the UK trial sites; plasma NEFL levels will be processed according to our previously published protocol

DETAILED DESCRIPTION:
In this proposed study we will use magnetic resonance imaging (MRI) of skeletal muscle to better delineate the natural history of intramuscular fat accumulation in Charcot Marie Tooth disease (CMT ) and investigate the use of muscle MRI and plasma neurofilament light chain (NEFL) levels as outcome measures in children and adults with specific subtypes of CMT (CMT1A, CMT1B, CMT2A and CMTX1).

We will ascertain the value of MRI-determined fat accumulation in foot, calf and thigh muscles as an independent outcome measure, by analysing its correlation with validated clinical measures [CMT Paediatric Score (CMTPedS) and/or CMT Examination Score version 2 - Rasch (CMTESv2-R)] and sensitivity to change over time compared to matched controls. We will also ascertain the utility of plasma NEFL levels as an independent outcome measure and a potential predictive biomarker of muscle fat accumulation over 12 months.

Following this trial, easily implemented outcome measures will be immediately available for clinical trials seeking to evaluate novel therapies in CMT and data from this trial will also be available to establish sample size for future clinical trials.

This study (participants with CMT and control participants) has two parts (Part 1: CMT1A cohort; Part2: CMT1B, CMT2A and CMTX1 cohort) and is proposed to take place over 3 years across three sites. Participants with CMT aged 5-60 for potential enrolment in the trial will be identified through the existing inherited neuropathy clinics at each site and control participants will be identified among the unaffected relatives and carers of the participants with CMT.

Approximately half of the participants will be recruited at the UK sites (NHNN and GOSH) and the other half at the US collaborating centre (University of IOWA). Each research visit is expected to last approximately 3 hours and during it, relevant detailed clinical data will be collected (CMTPedS for participants with CMT aged 5-20, CMTESv2-R for participants with CMT over the age of 10, CMT-HI for participants with CMT over the age of 16) and the participant will also undergo an MRI scan (up to 45 minutes) of the lower limbs (feet and calves or calves and thighs). Two separate neuromuscular MRI protocols with specific sequences will be used for the scans of foot and calf muscles and scans of calf and thigh muscles. Blood samples for plasma NEFL levels will be optional at both research visits for the participants at the UK trial sites; plasma NEFL levels will be processed according to our previously published protocol.

The primary objective is to define the responsiveness of MRI-determined fat accumulation in foot and calf muscles (in children/young adults aged 5-20 with CMT1A) or calf and thigh muscles (in adults aged 16-60 with CMT1B, CMT2A and CMTX1) over 12 months.

The secondary objectives are a) to assess the validity of MRI-determined muscle fat accumulation as a biomarker by correlating it with validated clinical scores (CMTPedS and/or CMTESv2-R), b) investigate the responsiveness of plasma NEFL in patients with CMT compared to matched controls over 12 months, and c) to investigate the utility of multi-level T2-weighted STIR (short T1 inversion recovery) and plasma NEFL levels as potential predictive biomarkers of muscle fat accumulation over the subsequent 12 months.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for participants with CMT

Part 1 inclusion criteria:

1. Participants aged 5-20 years with genetically proven CMT1A or with a clinical diagnosis of CMT1A (including neurophysiology) and a genetically confirmed diagnosis of CMT1A in patient or a 1st degree relative.
2. Participants must be able to undergo an MRI scan without sedation and complete the CMTESv2-R and/or CMTPedS scores as appropriate.
3. Female participants of childbearing potential who are sexually active must agree to use an effective method of contraception from the time consent is signed until the final research visit.
4. Female participants of childbearing potential must have a negative urinary pregnancy test prior to every MRI scan. Participants are considered not of childbearing potential if they are surgically sterile (i.e. they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal.
5. Participants and/or their parent(s)/guardian are willing and able to provide written informed consent and/or appropriate assent. Participants must have a good understanding of English language, in order to be able to do this.

Part 2 inclusion criteria:

1. Participants aged 16-60 years with genetically proven CMT1B, CMT2A or CMTX1 or with a clinical diagnosis of one of the above three (including neurophysiology) and a genetically confirmed diagnosis in a 1st degree relative.
2. Participants with CMTX1 must be male.
3. Participants must be able to undergo an MRI scan without sedation and complete the CMTESv2-R score.
4. Female participants of childbearing potential who are sexually active must agree to use an effective method of contraception from the time consent is signed until the final research visit.
5. Female participants of childbearing potential must have a negative urinary pregnancy test prior to every MRI scan. Participants are considered not of childbearing potential if they are surgically sterile (i.e. they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal.
6. Participants are willing and able to provide written informed consent. Participants must have a good understanding of English language, in order to be able to do this.

Inclusion criteria for control participants

1. Participants are aged 5-60 years.
2. Participants must be able to undergo an MRI scan without sedation.
3. Female participants of childbearing potential who are sexually active must agree to use an effective method of contraception from the time consent is signed until the final research visit.
4. Female participants of childbearing potential must have a negative urinary pregnancy test prior to every MRI scan. Participants are considered not of childbearing potential if they are surgically sterile (i.e. they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal.
5. Participants and/or their parent(s)/guardian are willing and able to provide written informed consent and/or appropriate assent. Participants must have a good understanding of English language, in order to be able to do this.

Exclusion Criteria:

Exclusion criteria for participants with CMT

1. Participants have undergone foot surgery in the 6 months prior to trial enrollment or are due to undergo foot surgery during the 12 months of the trial.
2. Participants have another medical condition which precludes them from having an MRI scan or completing the CMTESv2-R or the CMTPedS scores as appropriate.
3. Participants with known diagnosis of another neuromuscular disease.
4. Females who are planning pregnancy or breastfeeding

Exclusion criteria for control participants

1. Participants with known diagnosis of another neuromuscular disease.
2. A risk of developing a neuromuscular condition if the control participant is a relative of a participating patient with CMT.
3. Females who are planning pregnancy or breastfeeding

Ages: 5 Years to 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients aged 5-20 with genetically proven CMT1A, patients aged 16-60 with genetically proven CMT1B and CMT2A and male patients aged 16-60 with genetically proven CMTX1
Sampling Method: Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2018-09-11 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
MRI Change in fat accumulation in CMT1A | 12 months
  Part 1: Statistically significant (p<0.05) change of MRI-determined fat accumulation in foot and calf muscles in children/young adults with CMT1A over 12 months compared to matched controls.
MRI Change in fat accumulation in CMT1B; CMT2A and CMTX1 | 12 months
  Part 2: Statistically significant (p<0.05) change of MRI-determined fat accumulation in calf and thigh muscles in adults with CMT1B and CMT2A and male adults with CMTX1 over 12 months compared to matched controls.

SECONDARY OUTCOMES:
MRI changes validation - CMTPedS | 12 months
  Validating the change in MRI-determined fat accumulation in foot and calf muscles in children/young adults with CMT1A over 12 months by correlating it with the CMTPedS (all children) and the CMTESv2-R (children aged >10).
MRI changes validation - CMTESv2-R | 12 months
  Validating the change in MRI-determined fat accumulation in calf and thigh muscles in adults with CMT1B, CMT2A and CMTX1 over 12 months by correlating it with the CMTESv2-R
NEFL plasma responsiveness | 12 months
  Defining the responsiveness of plasma NEFL in patients with CMT compared to matched controls over 12 months.
NEFL plasma (biomarker) | 12 months
  Establishing the utility of plasma NEFL levels as a predictive biomarker of intramuscular fat accumulation over the subsequent 12 months in children/young adults with CMT1A.
Multi-level T2-weighted STIR and plasma NEFL levels (biomarker) | 12 months
  Establishing the utility of multi-level T2-weighted STIR and plasma NEFL levels as predictive biomarkers of intramuscular fat accumulation over the subsequent 12 months in adults with CMT1B, CMT2A and CMTX1

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Square Centre for Neuromuscular Diseases, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided